CLINICAL TRIAL: NCT05631847
Title: Endovascular Treatment With Or Without Intravenous Alteplase In Acute Ischemic Stroke Of Basilar Artery Occlusion: A Multicenter, Prospective, Randomized Controlled Trial (BEST-BAO)
Brief Title: Direct Endovascular Treatment Versus Bridging Treatment In Basilar Artery Occlusive Stroke
Acronym: BEST-BAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Academy of Medical Sciences (Other)
Collaborators: Sichuan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GFQ18981838913
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke; Basilar Artery Occlusion; Thrombosis; Alteplase; Endovascular Treatment
Keywords: Endovascular treatment; Alteplase; Acute ischemic stroke; Basilar artery occlusion; Intravenous thrombosis
MeSH Terms: conditions — Ischemic Stroke; Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct endovascular treatment group (Sham Comparator): Direct endovascular treatment (EVT) without intravenous thrombolysis (IVT)
  Interventions: Procedure: Endovascular treatment
- Bridging treatment group (Active Comparator): Intravenous thrombolysis (IVT) followed by endovascular treatment (EVT)
  Interventions: Procedure: Endovascular treatment; Drug: Intravenous thrombolysis (Alteplase)

INTERVENTIONS:
Procedure: Endovascular treatment — It is the emergency surgical removal of emboli which are blocking blood circulation. The strategies that were used for endovascular treatment included stent retrievers, thromboaspiration, balloon angioplasty, stent deployment, intraarterial thrombolysis (with alteplase), or combinations of these approaches that were left to the discretion of the treating team.
Drug: Intravenous thrombolysis (Alteplase) — Alteplase is used in the intravenous thrombolysis. It catalyzes the conversion of plasminogen to plasmin, the major enzyme responsible for clot breakdown.
  Arms: Bridging treatment group

SUMMARY:
Currently, both intravenous thrombolysis (IVT) followed by endovascular treatment (EVT) and EVT alone are widely used for the treatment of acute ischemic stroke (AIS) caused by basilar artery occlusion (BAO) (AIS-BAO), but no direct comparison of their efficacy and safety was reported. Only a limited number of cohort and registry studies have preliminarily compared the two strategies in the treatment of AIS-BAO, with results generally indicating that IVT followed by EVT was slightly superior to EVT alone. However, these findings are generally limited by small sample sizes, heterogeneous inclusion and exclusion criteria, different endpoint definitions, and distinct study designs, leading to inconsistent conclusions. Therefore, this study plans to conduct a multicentre, prospective, open-label, blinded endpoint evaluation, randomized controlled trial comparing the efficacy and safety of IVT followed by EVT and EVT alone in the treatment of patients with AIS-BAO who are eligible for both treatment strategies within 4.5 hours of symptom onset. This study intends to include patients with AIS due to BAO fulfilling the following inclusion criteria: patients with AIS caused by BAO confirmed by CTA/MRA/DSA; IVT can be started within 4.5 hours after symptoms onset; Age ≥ 18 years old; NIHSS score ≥ 6.

The primary endpoint of the study is the proportion of patients achieving mRS ≤ 2 at 90±14 days after stroke onset.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability in China, with acute ischemic stroke (AIS) accounting for approximately 85% of all acute strokes. Among these, large vessel occlusion-related AIS (AIS-LVO) represents about 20% of cases. Posterior circulation infarction, which occur in the vertebrobasilar artery territory, comprise 20-25% of all ischemic strokes. Although less common than anterior circulation ischemic strokes, posterior circulation infarctions-particularly AIS caused by basilar artery occlusion (AIS-BAO)-often present with severe symptoms and poor outcomes. Due to the heterogeneity of initial symptoms and diagnostic challenges, AIS-BAO frequently results in poor prognoses, posing significant challenges in clinical diagnosis and treatment.

The safety and efficacy of intravenous thrombolysis (IVT) with recombinant tissue plasminogen activator (rtPA) within 4.5 hours of symptom onset in AIS have been confirmed by numerous randomized controlled trials (RCTs). However, the heterogeneous presentation of posterior circulation AIS, the difficulty in clinical recognition compared to anterior circulation AIS, and the severe neurological deficits-especially the high mortality rate of AIS-BAO-pose various limitations on IVT. Endovascular treatment (EVT), including thrombectomy techniques, has substantially reduced the mortality and disability rates of patients with AIS-LVO. The key to treating AIS-BAO is recanalizing the acutely occluded basilar artery and rescuing the ischemic penumbra. Large RCTs have demonstrated that early EVT achieves better clinical outcomes in anterior circulation AIS-LVO patients eligible for mechanical thrombectomy compared to IVT alone.

In recent years, while multiple large RCTs have confirmed the efficacy of EVT for anterior circulation AIS-LVO, evidence for EVT in posterior circulation AIS-LVO remains limited. The BEST trial enrolled AIS patients with vertebrobasilar artery occlusion within 8 hours of symptom onset to compare EVT plus standard medical treatment versus medical treatment alone. The results showed that the combination group achieved better outcomes at 90 days, with no significant difference in mortality or symptomatic intracranial hemorrhage (sICH) rates compared to the medical treatment-only group. Similarly, the BASICS trial, an international multicenter RCT, enrolled 300 AIS-BAO patients within 6 hours of symptom onset and compared EVT combined with standard medical treatment to standard medical treatment alone. This study found no significant differences between the two groups in good functional outcomes, sICH, or mortality.

Recently, two studies focusing on thrombectomy for AIS-BAO reported promising results. The BAOCHE study randomized AIS-BAO patients who presented 6-24 hours after symptom onset into a thrombectomy plus standard medical treatment group or a standard medical treatment-only group. The primary endpoint was the proportion of patients with modified Rankin Scale (mRS) scores of 0-3 at 90 days. A total of 217 patients (110 in the combination group, 107 in the medical treatment group) were enrolled, and the results demonstrated that thrombectomy performed within 6-24 hours led to better functional outcomes at 90 days. The ATTENTION study, another RCT conducted across 36 stroke centers in China, enrolled AIS-BAO patients within 12 hours of symptom onset. Patients were randomized 2:1 to thrombectomy plus optimal medical treatment or optimal medical treatment alone. The primary outcome was the proportion of patients achieving an mRS score of 0-3 at 90 days, and 340 patients (226 in the combination group, 114 in the medical treatment group) were enrolled. The results showed that thrombectomy within 12 hours significantly improved functional outcomes. Both studies demonstrated that thrombectomy combined with medical treatment yielded better outcomes than medical treatment alone for AIS-BAO. However, questions remain regarding the optimal timing, treatment modalities, bridging strategies, and anesthesia options for EVT in posterior circulation AIS. Further exploration is required to rapidly identify posterior circulation strokes and select appropriate EVT strategies based on clinical indications.

Clinically, the morbidity and mortality of posterior circulation AIS-LVO exceed 80%. AIS-BAO, in particular, is a neurological emergency with extremely high mortality if untreated, significantly affecting patients' quality of life and imposing substantial medical and financial burdens on families and society. IVT remains the most effective ultra-early treatment for AIS within 6 hours of onset. However, the adoption of IVT for posterior circulation AIS is lower than that for anterior circulation AIS, potentially due to delays in diagnosis or missed diagnoses caused by the heterogeneity of AIS-BAO symptoms. Among AIS patients receiving IVT, posterior circulation strokes (PCS) account for about 5-19%. Studies comparing the efficacy and safety of IVT in PCS and anterior circulation strokes (ACS) have found that while the risk of hemorrhagic complications is halved for PCS, functional outcomes are similar, but mortality is higher. Clinically, IVT can be used as standalone therapy for AIS-BAO or as a prelude to EVT. Which approach better improves AIS-BAO outcomes remains uncertain.

To date, most studies on IVT with EVT have focused on anterior circulation AIS. Both IVT and EVT are time-dependent treatments for AIS, with EVT success hinging on prompt initiation and optimization of processes to reduce door-to-puncture time (DTP). The SKIP trial found no significant difference in the time from randomization to femoral artery puncture between only EVT and IVT with EVT. Similarly, the DEVT trial, conducted in China, also reported no difference in this time interval between the two groups. A meta-analysis of 38 observational studies including 11,798 AIS-LVO patients (56% of whom underwent IVT with EVT) also confirmed no significant difference in EVT procedural time between the two groups. For anterior circulation AIS-LVO, four recent RCTs showed mixed results. DIRECT-MT and DEVT demonstrated that only EVT was non-inferior to IVT with EVT in terms of good functional outcomes at 90 days, while SKIP and MR CLEAN-IV did not confirm non-inferiority. Thus, EVT alone requires further robust evidence[17, 18]. Regarding safety, all four RCTs confirmed that IVT with EVT does not increase sICH rates. Additionally, the aforementioned meta-analysis[16] confirmed that IVT with EVT does not increase sICH risk. SKIP, DIRECT-MT, and DEVT further showed no significant difference in mortality between the two groups. However, the meta-analysis suggested that IVT with EVT significantly reduces 90-day mortality compared to only EVT. A real-world study also found that IVT with EVT was independently associated with lower 90-day mortality compared to only EVT.

Does IVT before EVT achieve higher recanalization rates? A retrospective study including 93 AIS patients with middle cerebral artery occlusion showed that IVT with EVT resulted in a higher proportion of reperfusion within 1 hour of femoral artery puncture compared to only EVT. Moreover, IVT with EVT achieved significantly higher rates of successful reperfusion (mTICI ≥ 2b). The DIRECT-MT study found that IVT with EVT caused fewer new infarctions from thrombus fragmentation than only EVT. Similarly, post-hoc analyses of the ESCAPE trial demonstrated that IVT with EVT significantly reduced new infarct risk compared to only EVT. Another study of 57 patients with M1 segment occlusions reported that IVT with EVT often required fewer thrombectomy passes to achieve recanalization compared to only EVT.

Combination therapy combines the rapidity of IVT with the high recanalization rates of EVT, theoretically offering better outcomes than only EVT. However, most of these studies focus on anterior circulation stroke treatment. To date, no large-scale RCTs have specifically evaluated EVT with or without prior IVT for AIS-BAO. Therefore, we plan to conduct a multicenter, prospective, randomized controlled study to assess the impact of different EVT strategies on outcomes in AIS-BAO.

The primary objective of this trial is to compare the efficacy and safety of IVT followed by EVT versus EVT alone in patients with AIS caused by BAO who are eligible for both treatment strategies within 4.5 hours after symptom onset.

The secondary objectives include assessing the effects of the two treatment strategies on neurological function (assessed by National Institutes of Health Stroke Scale [NIHSS] score), activities of daily living (assessed by Barthel Index [BI] score), quality of life (assessed by EQ-5D-5L score), cerebrovascular reperfusion (assessed by eTICI), cerebrovascular recanalization (assessed by mAOL), infarct size (assessed by PC-ASPECTS and quantitative imaging detection), mortality, and the incidence of symptomatic intracranial hemorrhage (sICH).

This is a multicentre, prospective, open-label, blinded endpoint evaluation, randomized controlled clinical trial (PROBE design). Based on published observational studies, this trial will first validate the superiority of IVT followed by EVT compared with EVT alone. However, given the limited prior evidence and the current findings from anterior circulation stroke studies, this trial will also validate the non-inferiority of EVT compared with IVT followed by EVT alone if the efficacy of the two treatment strategies is found to be comparable.

An interim analysis is scheduled after one-third of the sample size completes follow-up for the primary endpoint. The primary purpose of the interim analysis is to allow for sample size re-estimation. The data and safety monitoring board (DSMB) will calculate the conditional power based on the current data and provide recommendations to the BEST-BAO research team regarding potential sample size adjustments.

The trial will be conducted at nationally recognized stroke centers and is expected to last for 3 years.

ELIGIBILITY:
Inclusion criteria:

1. A clinical diagnosis of AIS.
2. Caused by BAO confirmed by CTA, MRA, or DSA. (BAO is defined as the absence of visualization of the basilar artery on CTA, MRA or DSA. Bilateral vertebral artery occlusions or occlusion of a unilateral vertebral artery that is the sole supplier of the basilar artery, even in the presence of patent basilar artery, will be considered de facto BAO.)
3. CT or MRI ruling out intracranial hemorrhage,
4. Eligible for IVT and EVT (within 4.5 hours of symptom onset). (Symptoms onset is defined as point in time the patient was last seen well [at baseline] if patients are unable to provide a reliable history or the point in time when symptoms have started if patients can provide a reliable history. Symptoms onset includes diplopia, midline ataxia, visual loss, sensory or motor deficits, and conscious disturbance. Isolated vertigo [not accompanied by dysarthria, motor weakness, sensory symptoms, double vision, depressed level of consciousness] is not considered onset of symptoms.)
5. NIHSS score ≥ 6.
6. Age ≥ 18 years.
7. Signed informed consent by the patient or legal representative.

Exclusion criteria:

1. mRS score > 2 before this stroke.
2. Any contraindication to IVT as per the 2019 AHA/ASA guidelines for early management of AIS:

1) Blood pressure > 185/110 mmHg and cannot be controlled by standard medication, 2) Blood glucose < 50mg/dL (2.8 mmol/L) or > 400mg/dL (22.2 mmol/L), 3) Had a cerebral infarction in the previous 6 weeks with residual neurological deficit or signs of recent infarction on neuroimaging, 4) Severe head trauma in the previous 3 months, 5) Major surgery or severe trauma in the previous 2 weeks, 6) Gastrointestinal or urinary bleeding in the previous 3 weeks, 7) previous intracranial hemorrhage, 8) Using anticoagulants and International normalized ratio (INR) > 1.7, 9) Known platelet count < 100 × 109/L, 10) treatment with direct thrombin or factor X inhibitors, 11) Heparin treatment in the previous 48 hours with the activated partial thromboplastin time (APTT) exceeding the upper limit of normal.

(3) Pregnancy, breastfeeding, or intention to conceive during the study period. (4) Other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving mRS ≤ 2. | At 90±14 days after stroke onset.
  The mRS is an ordinal scale ranging from 0 to 6, where higher scores indicate a greater degree of disability.

SECONDARY OUTCOMES:
Proportions of patients with mRS = 0 or 1. | At 90±14 days after stroke onset.
  The mRS is an ordinal scale ranging from 0 to 6, where higher scores indicate a greater degree of disability.
Proportions of patients with mRS = 0-3. | At 90±14 days after stroke onset
  The mRS is an ordinal scale ranging from 0 to 6, where higher scores indicate a greater degree of disability.
The mRS score. | At 90±14 days after stroke onset
  The mRS score is an ordinal hierarchical scale ranging from 0 to 5, with higher scores suggesting more severe disability.
NIHSS (the National Institutes of Health Stroke Scale) score | At 18-24 hours after procedure, 24-74 hours after procedure, and 5-7 days after stroke onset and their changes from baseline.
  The NIHSS score is an ordinal hierarchical scale to evaluate the symptomatic severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores suggesting a more severe deficit.
Proportions of patients with a NIHSS score = 0 or 1, a NIHSS score = 0-2, a NIHSS score improvement ≥ 4 points, and a NIHSS score improvement ≥ 8 points. | At 18-24 hours after procedure, 24-74 hours after procedure, and 5-7 days after stroke onset.
  The NIHSS score is an ordinal hierarchical scale to evaluate the symptomatic severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores suggesting a more severe deficit.
Glasgow Coma Scale | At 18-24 hours after procedure, 24-74 hours after procedure, and 5-7 days after stroke onset and their changes from baseline.
  The Glasgow Coma Scale (GCS) is widely used to assess the level of consciousness in stroke patients, postoperative patients with brain injuries, and those with varying degrees of coma due to other causes.
BI score and the proportion with BI = 95-100. | At 30±7 and 90±14 days after stroke onset
  The Barthel Index (BI) is an ordinal scale used to measure performance in 10 activities of daily living. Scores range from 0 to 100, with higher scores indicating better performance in these activities.
EQ-5D-5L (the European Quality of Life 5-Dimension 5-Level) score | At 90±14 days after after stroke onset.
  The EQ-5D-5L score is an ordinal hierarchical scale to evaluate the quality of life. Scores range from -0.39 to 1, with higher scores indicating a better quality of life.
eTICI (Extended Treatment In Cerebral Ischemia) score and successful reperfusion rates. | Before and after EVT.
  The eTICI is an ordinal hierarchical scale ranging from 0 to 3, with higher scores suggesting better antegrade reperfusion of the previously occluded target artery ischemic territory.
mAOL score and recanalization rates | At 24-72 hours after procedure.
  The modified Arterial Occlusive Lesion (mAOL) scale is a standardized method used to evaluate arterial recanalization in acute ischemic stroke patients following endovascular treatment. It assesses the degree of reopening in the previously occluded artery, providing critical insights into the success of the intervention.
PC-ASPECTS score | At 24-72 hours after procedure and 5-7 days after stroke onset.
  The Posterior Circulation Alberta Stroke Program Early CT Score (PC-ASPECTS) is a standardized tool used to evaluate early ischemic changes in the posterior circulation territory.
Lesion volume. | At 24-72 hours after procedure and 5-7 days after stroke onset.
  Quantitative imaging detection.
All-cause mortality | Within 7, 30±7, and 90±14 days after stroke onset.
  The proportion of total deaths caused by various reasons in both arms
Proportions of patients with intracranial hemorrhage and symptomatic intracranial hemorrhage | At 24-72 hours after procedure and 5-7 days after stroke onset.
  The sICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 7 days or any hemorrhage leading to death.
New regional cerebral embolisms. | During EVT.
  Embolization to new territory assessment.Type A: Catheter was manipulated past the ostium of the new territory (e.g. large ACA infarct in a patient with an initial M1 occlusion): greater likelihood that infarct is related to the procedure.
  Type B: Catheter was not manipulated past the ostium of the new territory (e.g. left PICA infarct in a patient with an initial right M1 occlusion): lower likelihood that infarct is related to procedure.
Proportions of patients with new cerebral infarction | At 24-72 hours after procedure and 5-7 days after stroke onset.
  The proportion of the new cerebral infarction compared with the onset of symptoms evaluated with magnetic resource imaging test
EVT procedure-related complications. | Within 90±14 days after stroke onset.
  The pseudoaneurysm and hematoma at puncture site caused by various reasons is one of the important indicators reflecting puncture complications.

OTHER OUTCOMES:
Other serious adverse events. | Within 90±14 days after stroke onset.
  Other serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Qiang Guo, M.D., Principal Investigator — Sichuan Academy of Medical Sciences
Locations (96):
- China (96):
  - Banan Hospital Affiliated to Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Sanbo Chang'an Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Affiliated S Central Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Medical University Affiliated Yongchuan Hospital, Chongqing, Chongqing Municipality
  - Chongqing Yongchuan District People's Hospital, Chongqing, Chongqing Municipality
  - Hechuan District People's Hospital, Chongqing, Chongqing Municipality
  - Liangping District People's Hospital, Chongqing, Chongqing Municipality
  - The First People's Hospital of Liangjiang New Area, Chongqing, Chongqing Municipality
  - Zhangzhou Hospital, Zhangzhou, Fujian
  - The Fifth People's Hospital Affiliated to Southern Medical University, Guangzhou, Guangdong
  - Maoming County Traditional Chinese Medicine Hospital, Maoming, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Yulin First People's Hospital, Yulin, Guangxi
  - Qiandongnan Miao and Dong Autonomous Prefecture People's Hospital, Kaili, Guizhou
  - Anyang People's Hospital, Anyang, Henan
  - Jiaozuo Second People's Hospital, Jiaozuo, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Nanyang Nanshi Hospital, Nanyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Changde First People's Hospital, Changde, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Huai'an First People's Hospital, Huaian, Jiangsu
  - Jingjiang People's Hospital, Jingjiang, Jiangsu
  - The First People's Hospital of Suqian City, Suqian, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Xuzhou Medical University Affiliated Hospital, Xuzhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - Jilin University Sino Japanese Friendship Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Jilin, Jilin
  - Tieling Central Hospital, Tieling, Liaoning
  - Yingkou Central Hospital, Yingkou, Liaoning
  - Heze Municipal Hospital, Heze, Shandong
  - Liaocheng Second People's Hospital, Liaocheng, Shandong
  - Linyi Traditional Chinese Medicine Hospital, Linyi, Shandong
  - Rizhao Traditional Chinese Medicine Hospital, Rizhao, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Bazhong Central Hospital, Bazhong City, Sichuan
  - Chengdu Third People's Hospital, Chengde, Sichuan
  - Sichuan Third People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Chengdu First People's Hospital, Chengdu, Sichuan
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Chongzhou People's Hospital, Chengdu, Sichuan
  - Dayi County People's Hospital, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Western Theater General Hospital, Chengdu, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan
  - Shifang People's Hospital, Fangting, Sichuan
  - Guangyuan Central Hospital, Guangyuan, Sichuan
  - Guangyuan First People's Hospital, Guangyuan, Sichuan
  - Guang'an Central Hospital, Guang’an, Sichuan
  - Jintang County People's Hospital, Jintang, Sichuan
  - Leshan People's Hospital, Leshan, Sichuan
  - Guanghan People's Hospital, Luocheng, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Affiliated Traditional Chinese Medicine Hospital of Southwest Hospital Medical University, Luzhou, Sichuan
  - Meishan Cardiovascular and Cerebrovascular Disease Hospital, Meishan, Sichuan
  - Meishan Second People's Hospital, Meishan, Sichuan
  - Meishan Traditional Chinese Medicine Hospital, Meishan, Sichuan
  - Mianyang 404 Hospital, Mianyang, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Mianyang Third People's Hospital, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Langzhong People's Hospital, Nanchong, Sichuan
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Yilong County People's Hospital, Nanchong, Sichuan
  - Neijiang Second People's Hospital, Neijiang, Sichuan
  - Pangang Group General Hospital, Panzhihua, Sichuan
  - Panzhihua Central Hospital, Panzhihua, Sichuan
  - Pingchang County People's Hospital, Pingchang, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Suining First People's Hospital, Suining, Sichuan
  - Liangshan Prefecture Second People's Hospital, Xichang, Sichuan
  - Liangshan Prefecture First People's Hospital, Xichang, Sichuan
  - Ya'an People's Hospital, Ya'an, Sichuan
  - Yibin First People's Hospital, Yibin, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan
  - Zigong Fourth People's Hospital, Zigong, Sichuan
  - Zigong Third People's Hospital, Zigong, Sichuan
  - Lezhi County People's Hospital, Ziyang, Sichuan
  - Ziyang First People's Hospital, Ziyang, Sichuan
  - Qujing First People's Hospital, Qujing, Yunnan
  - Yongkang First People's Hospital, Guli, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiang Y, Yang S, Guo L, Dong C, Majoie CBLM, Siddiqui AH, Mocco J, Cavalcante F, Li BH, Wang JH, Huang B, Wang DZ, Yu NW, Schonewille WJ, Turk AS, Guo FQ. BEST-BAO: a multicentre, prospective, randomised controlled trial of endovascular treatment with or without intravenous thrombolysis in acute ischaemic stroke due to basilar artery occlusion - study protocol and rationale. Stroke Vasc Neurol. 2025 Oct 9:svn-2025-004144. doi: 10.1136/svn-2025-004144. Online ahead of print. PMID 40953924

DOCUMENTS (2):
  • Study Protocol (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT05631847/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT05631847/SAP_001.pdf